CLINICAL TRIAL: NCT03446716
Title: Effects of Sleep Extension on Sleep Physiology and Behavior of Young Children
Brief Title: Sleep Extension and Behavior of Young Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Rebecca Spencer, Associate Professor of Psychological and Brain Sciences, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-2739; R01HL111695 (NIH)
Record Dates: First submitted 2018-02-12; First posted 2018-02-27 (Actual); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Participants are assigned to the ADHD or Typically Developing group based on diagnosis history. Each then completes the intervention (EXTENSION) either preceded or followed by a week of baseline sleep (CONTROL). The order is pseudo-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EXTENSION (Experimental): During the extension condition, caregivers were instructed to put their child to bed 90 minutes earlier than their habitual bedtime for five consecutive nights. Caregivers were provided a list of tips to aid in implementing the earlier bedtime.
  Interventions: Behavioral: Sleep Extension
- CONTROL (No Intervention): Children followed their normal bedtime routine for five consecutive nights.

INTERVENTIONS:
Behavioral: Sleep Extension — Child attempted to go to bed 90 mins in advance of their normal bedtime.
  Arms: EXTENSION

SUMMARY:
This pseudo-randomized intervention study examined change in inhibitory control following a sleep manipulation in which children with and without ADHD were instructed to advance their bedtime by 90 minutes for five days.

DETAILED DESCRIPTION:
Objective: To evaluate the efficacy of a sleep extension intervention in young children with ADHD and determine whether sleep extension improves inhibitory control, a primary deficit in ADHD.

Design: Children with and without ADHD completed two 5-day assessments: a baseline condition in which children followed their normal bedtime routine and a sleep extension condition in which children were instructed to go to bed 90 minutes earlier than their habitual bedtime. Sleep was assessed with actigraphy and, on the final night, polysomnography. A Go/No-Go task was used to assess inhibitory control.

Setting: Participants slept in their home on nights 1-4 and in the sleep laboratory on night 5 of each condition.

Main Outcomes and Measures: Of interest is actigraph measurement of total sleep time for the baseline compared to the sleep extension condition. Polysomnography will be used to compared changes in sleep physiology. The primary behavioral outcome is inhibitory control, indexed by accuracy on No-Go trials in the Go/No-Go task.

ELIGIBILITY:
Inclusion Criteria:

* A subset of children were required to have an ADHD diagnosis

Exclusion Criteria:

* diagnosis of intellectual disabilities or developmental delay
* current diagnosis of history of sleep disorder
* uncorrected hearing or visual impairments

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 27 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2017-08-01 (Actual); Study Completion 2017-08-01 (Actual)

PRIMARY OUTCOMES:
total sleep time | 5 days (actigraph watch is worn for 5 days in each condition and overnight sleep time is identified and averaged across these 5 days)
  average nightly across 5 nights

SECONDARY OUTCOMES:
inhibitory control | measured before and after sleep - about 12 hrs
  measured with the Go/NoGo task

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Spencer, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (1):
- University of Massachusetts, Amherst, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-20): https://cdn.clinicaltrials.gov/large-docs/16/NCT03446716/Prot_SAP_000.pdf